CLINICAL TRIAL: NCT04819451
Title: Effect of Magnesium-rich Artificial Cerebrospinal Fluid Replacement on the Prognosis of Patients With Subarachnoid Hemorrhage
Brief Title: Application of Magnesium-rich Artificial Cerebrospinal Fluid in Subarachnoid Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XJTU1AF2020LSK-195
Record Dates: First submitted 2021-03-09; First posted 2021-03-29 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Intracranial Hemorrhage
Keywords: Intracranial Hemorrhage; Artificial cerebrospinal fluid; Cerebrospinal fluid replacement; Subarachnoid Hemorrhage
MeSH Terms: conditions — Intracranial Hemorrhages; Subarachnoid Hemorrhage

STUDY DESIGN:
Intervention Model Description: rospective, interventional, double-blind, completely randomized, stratified controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MACSF group (Experimental): In the experimental group, patients with intracerebral hemorrhage ruptured into the ventricle and patients with subarachnoid hemorrhage were included in the stratified random method. Use Magnesium-Rich Artificial Cerebrospinal Fluid(MACSF) in the CSF replacement, and the remaining treatments should strictly follow the guidelines as same as the control group. The total amount of replacement was generally 30ml, and the replacement was performed once every 3 days. When the RBC count in CSF is less than 100×10^6/L, the CSF is considered to be cleared. Cerebrospinal fluid replacement is performed up to four times.
  Interventions: Other: Magnesium-Rich Artificial Cerebrospinal Fluid (MACSF)
- NS group (No Intervention): In the control group, patients with intracerebral hemorrhage ruptured into the ventricle and patients with subarachnoid hemorrhage were included according to the stratified random method. Use the normal saline (0.9% Sodium Chloride Injection) in the CSF replacement, and the remaining treatments should strictly follow the guidelines. The total amount of replacement was generally 30ml, and the replacement was performed once every 3 days. When the RBC count in CSF is less than 100×10^6/L, the CSF is considered to be cleared. Cerebrospinal fluid replacement is performed up to four times.

INTERVENTIONS:
Other: Magnesium-Rich Artificial Cerebrospinal Fluid (MACSF) — The Magnesium-Rich Artificial Cerebrospinal Fluid (MACSF) is composed of several qualified clinical intravenous injections according to a specific formula, which has similar physical and chemical properties to physiological CSF. MACSF will be freshly made and used. It will be prepared by trained professionals on a specific workbench and sent to the patient wards in a special container. Finally, it will be used in the CSF replacement. Aseptic principles should be enforced strictly during the whole procedures, including preparation, transportation and application.
  Arms: MACSF group

SUMMARY:
Intracerebral hemorrhage (ICH) is one of the common fatal types of cerebral apoplexy with high mortality and disability rates. Hematoma volume and complications of intracerebral hemorrhage are major predictors of early death and poor prognosis. The hematoma and its metabolites are key therapeutic targets. At present, in order to improve the prognosis of patients, cerebrospinal fluid(CSF) replacement with normal saline(NS) is commonly used in clinical practice to clear the bloody components, which shows a good clinical effect. However, due to the large difference between NS and CSF composition, it is easy to cause secondary injury of brain tissue. Therefore, the replacement of artificial CSF with similar CSF composition will be more effective in reducing the incidence of complications and improve the prognosis of neurological function.

The Magnesium-rich Artificial Cerebrospinal Fluid(MACSF) was designed and developed in the early stage of this project which has similar physical and chemical properties to physiological CSF, such as ion species, concentration, the potential of hydrogen (pH) value, and osmotic pressure. Animal experiments had confirmed its safety and effectiveness. In this study, patients with basal ganglia intracerebral hemorrhage ruptured into the ventricle or subarachnoid hemorrhage were stratified randomly divided into MACSF group and NS group. MACSF and NS were used as replacement fluid for lumbar puncture CSF replacement, respectively. By observing and comparing two groups of patients of the Modified Rankin Scale (mRS) on the days14, 30, 60 and 90 after onset; hematoma absorption rate, hemorrhagic CSF removal rate; changes of cerebral autoregulation； incidence of complications, such as acute obstructive hydrocephalus (AOH) and cerebral vasospasm (CVS); the changes of scores and scales about imaging; assessment of neurological function recovery, such as the National Institutes of Health Stroke Scale (NIHSS) and the Glasgow Coma Score (GCS) during hospitalization, headache duration and the Visual Analogue Scale (VAS), vomiting duration, duration of meningeal irritant, ICU hospitalization duration, total hospitalization duration; change of CSF and peripheral blood biochemical indicators. The objective is to evaluate MACSF replacement therapy in patients with basal ganglia cerebral hemorrhage broken into ventricles and nonaneurysmal subarachnoid hemorrhage of the influence of absorption rate and prognosis.

DETAILED DESCRIPTION:
This study is a prospective, interventional and double-blind randomized controlled clinical trial. After approval of the clinical registry, patients who meet the standards of inclusion and exclusion criteria will be recruited to this study, if they and their relatives are willing to join the study. According to the clinical manifestations of the patients at admission and the results of cranial imaging, the patients' conditions were evaluated using the modified Fisher score, the World Federation of Neurological Surgeons Scale (WFNSS), the max-ICH score (max-ICH), the IVH score (IVHs), the Hijdra Sum Score (Hijdra), the Modified Graeb Score (mGS) and other grading criteria. Two groups (NS group and MACSF group) were divided into groups using a completely stratified randomization method. This study was a double-blind clinical study, and the grouping protocol was managed by the project research assistant. After the subject or his/her family members sign the informed consent, the project research assistant completed the grouping according to the randomly assigned sequence given by the clinical research center of the First Affiliated Hospital of Xi'an Jiaotong University. The project research assistant records the group and informs the specialist of the type of replacement fluid required. The replacement fluid was sent into the ward in a special container, and then lumbar puncture and CSF replacement were performed by the operator. The replacement liquid used in both groups was identical in appearance, color, temperature, and smell. During the whole study, the investigator did not participate in the preparation of the replacement liquid, and the subjects and their family members were also unaware of the grouping. After the case collection and electronic database records are completed, the research assistant will inform the researcher of the group name under the supervision of the third party to complete the unblinding, and the researcher shall inform the subjects of the group name in written form. For the control group, patients have treated the normal saline (0.9% Sodium Chloride Injection) as the replacement fluid. For the intervention group, MACSF will be used. The composition and concentration of MACSF is as follows:Na+: 146.2 mEq/L, K+: 2.7 mEq/L, Mg2+: 4.2 mEq/L, Cl-: 123 mEq/L, HCO3-:23.2 mEq/L, Glucose: 0.75 g/L. MACSF is prepared by the Pharmacy Intravenous Admixture Services staff of First Affiliated Hospital of Xi'an Jiaotong University, according to a specific formula in the specific working area. The whole procedure follows the aseptic principles strictly. Fresh-made MACSF will be placed in a specific container and sent to the patient ward through specific channels. Intracranial pressure (ICP) was measured by a non-invasive ICP test before lumbar puncture. If it is higher than 350cmH2O, a lumbar puncture can be performed 30 minutes after an intravenous drip of 100ml 20% mannitol. Then, for the patients who signed the informed consent, a CSF sample (3ml) was taken before each lumbar puncture CSF replacement and synchronous blood samples (6ml) were taken. The blood samples should be drawn into a non-anticoagulant tube and a heparin anticoagulant tube respectively. All the samples will be transferred to BioBank of the First Affiliated Hospital of Xi'an Jiaotong University in a liquid nitrogen tank. After re-melted in a water bath of 37°, the blood samples will be centrifuged at 4° for 15min at 3000r/min, the CSF samples will be centrifuged at 4° for 10min at 1000r/min and then the supernatant will be collected and stored at -80°. At the end of this study, the contents of oxyhemoglobin (oxy-Hb), S100 calcium-binding protein β (S100β), neuron-specific enolase(NSE), D-dimer (DD), matrix metalloproteinases-9 (MMP-9), Mg2+, Ca2+ in the samples will be detected by enzyme-linked immunosorbent assay (ELISA) or mass spectrometry. The total amount of replacement was generally 30ml, and the replacement was performed once every 2 days. When the red cell (RBC) count in CSF is less than 100×10^6/L, the CSF is considered to be cleared. CSF replacement is performed up to four times. NIHSS and GCS scores were evaluated daily after admission. Cerebral computerized tomography (CT) was performed at least every week after admission. If there are new low-density lesions, delayed cerebral infarction (DCI) will be diagnosed. A transcranial Doppler(TCD) examination was performed the first three days after admission and after each replacement. Cerebral autoregulation (CA) was evaluated by transient hyperemic response test (THRT), a transcranial Doppler (TCD)-based CA evaluation method, which describes the changes in cerebral blood fow velocity after a brief compression of the ipsilateral common carotid artery. The specific content is described later. CVS will be diagnosed by TCD, the diagnostic criteria will be described later. All subjects were followed up on the 14, 30, 60, and 90 days after onset, and the mRS was evaluated. Meanwhile, some indicators will be used to evaluate the safety of MACSF application, which include secondary infection, fluctuation of intracranial pressure, and hypermagnesemia. For patients or their family members who do not agree to do the CSF replacement, the sample collection can be used as a supplementary analysis for this study after they sign the informed consent for sample collection.

The diagnostic criteria and the solutions will be described in the next part.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 18 and 80 years of old;
* Patients with ICH rupture into the ventricle in the primary basal ganglia region or non-aneurysmal subarachnoid hemorrhage confirmed by skull imaging examination;
* Patient is admitted to hospital within 72 hours after onset;
* Informed consent of the patients or their family members, and signed informed consent for CSF replacement treatment.

Exclusion Criteria:

* Non-spontaneous intracranial hemorrhage;
* Time from onset to admission is longer than 72 hours;
* The patient who needs surgical treatment;
* Contraindication of lumbar puncture, such as: cerebral hernia, severe intracranial hypertension, puncture site inflammation, blood system diseases, etc.;
* Patient has other serious diseases, such as heart failure, kidney failure, liver failure, etc;
* Patient or his/her relatives refuse to accept the above research plan.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
The mRS score at 14, 30, 60,90 days after onset | in the day of 14, 30, 60, 90 days after onset.
  Assess patients' prognosis by the score of modified Rankin Scale.In the mRS, the lowest score is 0, and the highest score is 5. A score of 0 indicates the patients have no symptoms at all, and a score of 5 indicates the patients have severe disability, bed rest, incontinence, and need for continuous care and attention. In this study, we evaluate patient's outcomes by the following criteria. Favorable outcome was defined as mRS<3, whereas poor outcome was mRS≥3.

SECONDARY OUTCOMES:
Clearance rate of hemorrhagic CSF | Within 30 days after onset.
  Record the number of days from the first CSF replacement to the end of replacement and the red blood cell count in CSF. The difference of CSF red blood cell count was divided by the number of days to calculate the clearance rate of hemorrhagic CSF.
The absorption rate of hematoma | Within 30 days after onset.
  The absorption rate of hematoma (ml/d)=(the volume of the first CT hematoma-the volume of the other CT hematoma after the replacement)/ the interval time;Total hematoma volume (TV)=ICH volume +IVH volume;ICH volume =ABC/2; Method: where A is the longest diameter of the largest hematoma layer on CT,B is the longest diameter perpendicular to line A, and C is the thickness of the visible layer of the hematoma = the number of layers of scan spacing];IVH volume was calculated by IVH score/ Graeb score.
CT imaging: The max-ICH score (max-ICH) | Within 30 days after onset.
  The minimum value is 0 and maximum value is 10, and higher scores mean a worse outcome.
CT imaging: the IVH score (IVHs) | Within 30 days after onset.
  The minimum value is 0 and maximum value is 9, and higher scores mean a worse outcome.
CT imaging: the Modified Graeb Score (mGS) | Within 30 days after onset.
  The minimum value is 0 and maximum value is 32, and higher scores mean a worse outcome.
CT imaging: the Hijdra Sum Score (Hijdra) | Within 30 days after onset.
  The minimum value is 0 and maximum value is 27, and higher scores mean a worse outcome.
Incidence and severity of cerebral vasospasm(CVS) | Within 20 days after onset.
  Transcranial Doppler (TCD) will be used to evaluate the occurrence and severity of CVS, which will be diagnosed according to the following criteria for TCD. First, the mean blood flow velocity of tested arteries is higher than 120cm/ s. Second, the mean blood flow velocity of tested arteries increases more than 15cm/s or 20% compared with the previous time. Third, the Lindeggard Index (mean blood flow velocity of middle cerebral artery/mean blood flow velocity of ipsilateral eICA) is higher than 3. TCD was performed within 72 hours after onset and after each cerebrospinal fluid replacement.
Changes in cerebral autoregulation (CA) | Within 20 days after onset.
  CA was evaluated by transient hyperemic response test (THRT), a transcranial Doppler (TCD)-based CA evaluation method, which describes the changes in cerebral blood fow velocity after a brief compression of the ipsilateral common carotid artery. Transient hyperemic response ratio (THRR) to the baseline blood flow velocity (the mean of the blood flow velocity in the first five systolic periods of compression) was calculated, which reflected the automatic regulation function of cerebral blood flow after hyperperfusion. Bilateral THRR≥1.09 is considered to have normal automatic regulation function, unilateral THRR≤1.09 considers that the function of automatic regulation is impaired. TCD was performed within 72 hours after onset and after each cerebrospinal fluid replacement.
Incidence and severity of acute obstructive hydrocephalus(AOH) | Within 20 days after onset.
  For included patients, the size of the ventricular system will be measured by means of calculating the bicaudate index(BCI): "The width of the frontal horns at the level of the caudate nuclei divided by the corresponding diameter of the brain." The relative BCI was obtained by dividing the patient's BCI by the normal upper limit (95th percentile) for age. Acute hydrocephalus was defined as a relative BCI of more than one.
Incidence of the second stroke and the mortality | Within 90 days after onset.
  Stroke was determined by CT or MRI and mortality was recorded.
Neurological function recovery | Within 20 days after onset.
  The National Institutes of Health Stroke Scale (NIHSS) and the Glasgow Coma Score (GCS) score during hospitalization. The value of NIHSS is 0 to 34, and higher scores mean a worse outcome. The value of GCS is 0 to 16, and higher scores mean a better outcome.
Differences in duration of neurological symptoms | Within 20 days after onset.
  Record the headache duration (day) and the Visual Analogue Scale (VAS), duration and dosage of analgesics, vomiting duration (day), duration of meningeal irritant (day). The minimum value of the Visual Analogue Scale (VAS) is 0 and maximum value is 100, and higher scores mean a worse outcome.
Duration of hospitalization | Within 60 days after onset.
  ICU hospitalization duration (day), total hospitalization duration (day).
Levels of biomarkers in cerebrospinal fluid(CSF) and blood | Within 20 days after onset.
  For the patients who signed the informed consent, a CSF sample (3ml) was taken before each lumbar puncture CSF replacement and synchronous blood samples (6ml) was taken to evaluate the effect of MACSF on oxyhemoglobin(OxyHb, ng/L), S100 calcium-binding protein β(S100β, ng/L), neuron-specific enolase(NSE, ng/L), D-dimer(DD, ng/L), matrix metalloproteinases(MMPs, ng/L).
Levels of ion concentration in CSF and blood | Within 20 days after onset.
  For the patients who signed the informed consent, a CSF sample (3ml) was taken before each lumbar puncture CSF replacement and synchronous blood samples (6ml) was taken to evaluate the effect of MACSF on Mg2+ (mEq/L)and Ca2+ (mEq/L).

OTHER OUTCOMES:
Fluctuation of intracranial pressure(ICP) | Before each cerebrospinal fluid replacement during the hospitalization.
  ICP will be assessed by non-invasive ICP monitoring and lumbar puncture. The severity will be evaluated by days of use of dehydrated drugs.
Incidence and severity of MACSF-induced infection | Within 20 days after onset.
  If the patient has some symptoms of infection, the doctor in charge must determine whether it is MACSF-induced infection and assess the severity. First, the MACSF-induced infection will be diagnosed by the patient's symptoms and the MACSF sample's pathogenic detection. Second, the severity of infection will be evaluated by the indicators including the duration of fever, the kinds of antibiotics, the duration of antibiotics use and the results of CSF examination.
Incidence of hypermagnesemia | Within 20 days after onset.
  Pay close attention to the clinical manifestations of fatigue, disappearance of tendon reflex and decreased blood pressure, and monitor the blood electrolyte level dynamically to assess the incidence of hypermagnesemia.

CONTACTS AND LOCATIONS:
Overall Officials: Guogang Luo, MD, PHD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes